CLINICAL TRIAL: NCT02732600
Title: Program Evaluation of Peer Specialists on VA PACTS: A Quality Improvement Project (QUE 15-289)
Brief Title: Evaluation of Peer Specialists on VA PACTs
Acronym: Peers on PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: QUX 16-001
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Results first posted 2020-06-12 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Mental Illness; Physical Illness
Keywords: Veterans; Veterans Health; Patient Compliance; Primary Health Care; Health Care Providers; Health Promotion
MeSH Terms: conditions — Mental Disorders; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Implementation (No Intervention): Standard Implementation sites will receive written guidance and limited consultation by the investigators' team.
- Facilitated Implementation (Experimental): Facilitated Implementation sites will receive one year of support based on the i-PARIHS implementation model which includes training, implementation planning, ongoing external facilitation, feedback and consultation.
  Interventions: Other: Facilitated Implementation

INTERVENTIONS:
Other: Facilitated Implementation — Facilitated Implementation sites will receive one year of support based on the i-PARIHS implementation model which includes training, implementation planning, ongoing external facilitation, feedback and consultation
  Arms: Facilitated Implementation

SUMMARY:
In August 2014, the White House issued an Executive Action mandating that 25 VA medical centers place Peer Specialists (Veterans recovered from mental illness who are trained to support other Veterans with mental illness) on Primary Care Teams. Research shows that the success of adding new staff to existing teams can be improved by outside aid and facilitation. This quality improvement project will evaluate whether providing expanded support to half of the Primary Care Teams will lead to better outcomes when compared with teams that do not get extra support.

DETAILED DESCRIPTION:
Peer Specialists are individuals with mental illness currently deployed to serve Veterans in specialty mental health clinics based upon their lived experiences. Peer Specialist delivered interventions have been shown to improve patient activation in multiple studies. In August 2014, the White House issued an Executive Action mandating that 25 VA medical centers pilot the deployment of Peer Specialists in their Patient Aligned Care Teams (PACTs). This project expands upon this nationally mandated Peer Specialist pilot with the integration of a cluster randomized implementation trial. This quality improvement project will evaluate the impact of facilitated implementation vs. standard implementation to support on the deployment of Peer Specialists in PACTs.

The 25 sites will be divided into three cohorts (n=8,8,9). Each cohort will begin over three successive six-month blocks beginning in early 2016. Within each cohort, sites will be randomized to receive either facilitated or standard implementation. Facilitated Implementation sites will receive one year of support based on the i-PARIHS implementation model which includes training, implementation planning, ongoing external facilitation, feedback and consultation. Standard Implementation sites will receive written guidance and limited consultation by the investigators' team. The investigators will compare the groups on 1) the percent of their target population that actually received PS services; 2) ratings on PS workload productivity including ; 3) Peer Implementation and Services scores; 4) assessment of Veteran's change over time on the outcome variables of satisfaction, activation, and functioning ; 5) qualitative analysis of how well PSs were deployed and their impact.

ELIGIBILITY:
Inclusion Criteria:

* Included sites must be VA PACT Primary Care Health teams with existing Peer Specialists who are able to include an existing Peer Specialist on their team for a minimum of 10 hours per week for one year

Exclusion Criteria:

* Non VA PACT teams, VA sites without an existing Peer Specialists, and VA PACT primary care teams that cannot commit a Peer Specialist to Primary Care for a minimum of 10 hours per week are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5616 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Chinman, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA; Richard W Goldberg, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (25):
- United States (25):
  - Southern Arizona VA Health Care System, Tucson, AZ, Tucson, Arizona
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - West Palm Beach VA Medical Center, West Palm Beach, FL, West Palm Beach, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - VA Northern Indiana Health Care System Marion Campus, Marion, IN, Marion, Indiana
  - Lexington VA Medical Center, Lexington, KY, Lexington, Kentucky
  - Maine VA Medical Center, Augusta, ME, Togus, Maine
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts
  - John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York
  - Salisbury W.G. (Bill) Hefner VA Medical Center, Salisbury, NC, Salisbury, North Carolina
  - Chillicothe VA Medical Center, Chillicothe, OH, Chillicothe, Ohio
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - Chalmers P. Wylie Ambulatory Care Center, Columbus, OH, Columbus, Ohio
  - Philadelphia VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Wm. Jennings Bryan Dorn VA Medical Center, Columbia, SC, Columbia, South Carolina
  - White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peeples AD, Muralidharan A, McCarthy S, Goldberg R, Kuykendall L, Vineyard N, Chinman M. Barriers and Enablers to Implementing Peer Specialists in Veterans Health Administration Primary Care: a Qualitative Study. J Gen Intern Med. 2023 Feb;38(3):707-714. doi: 10.1007/s11606-022-07782-0. Epub 2022 Sep 20. PMID 36127539
- [Derived] Chinman M, Goldberg R, Daniels K, Muralidharan A, Smith J, McCarthy S, Medoff D, Peeples A, Kuykendall L, Vineyard N, Li L. Implementation of peer specialist services in VA primary care: a cluster randomized trial on the impact of external facilitation. Implement Sci. 2021 Jun 7;16(1):60. doi: 10.1186/s13012-021-01130-2. PMID 34099004
- [Derived] Chinman M, Daniels K, Smith J, McCarthy S, Medoff D, Peeples A, Goldberg R. Provision of peer specialist services in VA patient aligned care teams: protocol for testing a cluster randomized implementation trial. Implement Sci. 2017 May 2;12(1):57. doi: 10.1186/s13012-017-0587-7. PMID 28464935

RESULTS

PARTICIPANT FLOW:
Recruitment Details: numbers of participants is presented at three time points: 1. Baseline 2. 6-months, and 3. 1-year
Units Other Than Participants: Sites
Period: Overall Study
Arm/Group | Standard Implementation | Facilitated Implementation
Started | 3525; 13 Sites | 2091; 12 Sites
Sub-set of Sites Newly Delivering PS Services | 899; 12 Sites | 1484; 11 Sites
Veteran Baseline Veteran (Sub-set of 23 Sites) | 118; 12 Sites | 145; 11 Sites
Veteran 6-months (Sub-set 23 Sites) | 70; 12 Sites | 84; 11 Sites
Veteran 1-year (Sub-set 23 Sites) | 54; 12 Sites | 71; 11 Sites
Peer Specialist Responses at 6-months (All 25 Sites) | 12; 13 Sites | 14; 12 Sites
Peer Specialist Responses at 1-year (All 25 Sites) | 5; 13 Sites | 12; 12 Sites
Supervisor Responses 6-months (All 25 Sites) | 10; 13 Sites | 21; 12 Sites
Supervisor 1-year (All 25 Sites) | 6; 13 Sites | 10; 12 Sites
Completed (These are the number of Veterans (across all 25 sites) who completed surveys) | 100; 13 Sites | 113; 12 Sites
Not Completed | 3425; 0 Sites | 1978; 0 Sites

BASELINE CHARACTERISTICS:
Population: baseline characteristics only completed for Veterans completing surveys
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Implementation | Facilitated Implementation | Total
Number analyzed (Participants) | 194 | 221 | 415
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: numbers vary across variables due to missing data
  years
    number analyzed (Participants) | 160 | 208 | 368
    (all) | 61.1 (10.7) | 61.2 (13.8) | 61.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants] — numbers vary from total sample due to missing data Population: numbers vary from total due to missing data
  Participants
    number analyzed (Participants) | 160 | 203 | 363
    Female | 28 | 17 | 45
    Male | 132 | 186 | 318
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: numbers vary due to missing data
  Participants
    number analyzed (Participants) | 152 | 196 | 348
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 37 | 64 | 101
    White | 109 | 121 | 230
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 6 | 11 | 17

OUTCOME MEASURES:

1. Primary Outcome: Patient Activation Measure Change
Description: The Patient Activation Measure (PAM) is a 13-item survey that measures an individual's perceived ability to manage his or her illness and health behaviors and act as an effective patient. It has been shown to be reliable, valid, sensitive to change and correlates with measures of improved self-management. Scores for this outcome range from Zero to One Hundred with higher scores indicating higher levels of patient activation (better outcome).
Time Frame: Baseline, 6 months, 1 year
Population: Comparison across two conditions on PAM Total Score - PAM Total Score (0-100)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Standard Implementation | Facilitated Implementation
Number analyzed (Participants) | 194 | 221
Score on a scale
  Baseline-PAM Total | 41.0 (5.9) | 41.6 (6.2)
  6-Month-PAM Total: number analyzed (Participants) | 121 | 129
  6-Month-PAM Total | 39.9 (5.6) | 40.6 (5.7)
  1-year-PAM Total: number analyzed (Participants) | 100 | 113
  1-year-PAM Total | 39.8 (6.2) | 40.8 (5.5)
Statistical Analysis 1: Comparison: Standard Implementation vs Facilitated Implementation; Analysis 1 is Comparison Across Conditions at BASELINE Analysis 2 is Comparison Across Conditions at 6 Months Analysis 3 is Comparison Across Conditions at 1 year; Test type: Superiority; p = 0.39, t-test, 2 sided; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [-0.66 to 1.68], Standard Error of Mean 0.59
Statistical Analysis 2: Comparison: Standard Implementation vs Facilitated Implementation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.35, t-test, 2 sided; Mean Difference (Final Values) = 0.65, 95% CI 2-sided [-0.75 to 2.06], Standard Error of Mean 0.71
Statistical Analysis 3: Comparison: Standard Implementation vs Facilitated Implementation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.21, t-test, 2 sided; Mean Difference (Final Values) = 1.01, 95% CI 2-sided [-0.57 to 2.60], Standard Error of Mean 0.81

2. Secondary Outcome: Team Development Measure
Description: The Team Development Measure is a 31 item self-report survey that evaluates the degree to which a team has and uses the components needed for highly effective teamwork including cohesiveness, communication, role clarity, and goals and means clarity. All components min scores are zero % and maximum is 100%; higher percentages mean positive responses.
Time Frame: Baseline, 6 months, 1 year
Population: number of site based leadership and supervisors who responded
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Implementation | Facilitated Implementation
Number analyzed (Participants) | 21 | 30
units on a scale
  cohesiveness-Baseline | 91.1 (15.5) | 96.7 (10.3)
  Communication Baseline | 85.0 (22.4) | 93.0 (19.5)
  Role Clarity Baseline | 76.0 (28.6) | 84.4 (16.3)
  Goals Baseline: number analyzed (Participants) | 21 | 20
  Goals Baseline | 67.9 (38.9) | 82.0 (29.9)
  Cohesiveness 6 month: number analyzed (Participants) | 21 | 20
  Cohesiveness 6 month | 89.6 (21.8) | 89.1 (23.5)
  Communication 6 month: number analyzed (Participants) | 21 | 20
  Communication 6 month | 84.7 (26.9) | 86.0 (26.9)
  Role Clarity 6 months: number analyzed (Participants) | 21 | 20
  Role Clarity 6 months | 77.0 (31.8) | 83.2 (22.3)
  Goals 6 months: number analyzed (Participants) | 21 | 20
  Goals 6 months | 74.8 (28.6) | 77.0 (19.8)
  Cohesiveness 1 year: number analyzed (Participants) | 8 | 16
  Cohesiveness 1 year | 85.2 (35.0) | 94.3 (13.2)
  Communication 1 year: number analyzed (Participants) | 8 | 16
  Communication 1 year | 80.0 (32.1) | 83.2 (22.9)
  Role Clarity 1 year: number analyzed (Participants) | 8 | 16
  Role Clarity 1 year | 70.8 (40.6) | 82.3 (21.5)
  Goals 1 year: number analyzed (Participants) | 8 | 16
  Goals 1 year | 77.5 (24.9) | 87.5 (17.7)
Statistical Analysis 1: Comparison: Standard Implementation vs Facilitated Implementation; t-test used to compare group differences in Cohesiveness at BASELINE; Test type: Superiority; p = 0.156, t-test, 2 sided; Mean Difference (Final Values) = 5.61, 95% CI 2-sided [-2.2 to 13.48], Standard Error of Mean 3.6
Statistical Analysis 2: Comparison: Standard Implementation vs Facilitated Implementation; t-test to compare group means on Communication at BASELINE; Test type: Superiority; p = 0.182, t-test, 2 sided; Mean Difference (Final Values) = 7.97, 95% CI 2-sided [-3.85 to 19.8], Standard Error of Mean 5.89
Statistical Analysis 3: Comparison: Standard Implementation vs Facilitated Implementation; t-test to compare group differences on Role Clarity at BASELINE; Test type: Superiority; p = 0.234, t-test, 2 sided; Mean Difference (Final Values) = 8.41, 95% CI 2-sided [-5.74 to 22.57], Standard Error of Mean 6.31
Statistical Analysis 4: Comparison: Standard Implementation vs Facilitated Implementation; t-test to compare group values on Goals at Baseline; Test type: Superiority; p = 0.149, t-test, 2 sided; Mean Difference (Final Values) = 14.14, 95% CI 2-sided [-5.22 to 33.5], Standard Error of Mean 9.63
Statistical Analysis 5: Comparison: Standard Implementation vs Facilitated Implementation; t-test of differences between groups on Cohesiveness at 6-Months; Test type: Superiority; p = 0.947, t-test, 2 sided; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-14.7 to 13.8], Standard Error of Mean 7.1
Statistical Analysis 6: Comparison: Standard Implementation vs Facilitated Implementation; t-test of groups differences on Communication at 6 Months; Test type: Superiority; p = 0.870, t-test, 2 sided; Mean Difference (Final Values) = 1.38, 95% CI 2-sided [-15.6 to 18.4], Standard Error of Mean 8.4
Statistical Analysis 7: Comparison: Standard Implementation vs Facilitated Implementation; t-test of group differences on Role Clarity at 6 months; Test type: Superiority; p = 0.478, t-test, 2 sided; Mean Difference (Final Values) = 6.18, 95% CI 2-sided [-11.26 to 23.63], Standard Error of Mean 8.62
Statistical Analysis 8: Comparison: Standard Implementation vs Facilitated Implementation; t-test of group differences on Goals at 6 Months; Test type: Superiority; p = 0.773, t-test, 2 sided; Mean Difference (Final Values) = 2.23, 95% CI 2-sided [-13.35 to 17.83], Standard Error of Mean 7.71
Statistical Analysis 9: Comparison: Standard Implementation vs Facilitated Implementation; t-test of group differences on Cohesiveness at 1year; Test type: Superiority; p = 0.498, t-test, 2 sided; Mean Difference (Final Values) = 9.09, 95% CI 2-sided [-20.4 to 38.6], Standard Error of Mean 9.8
Statistical Analysis 10: Comparison: Standard Implementation vs Facilitated Implementation; t-test of group differences on Communication at 1 year; Test type: Superiority; p = 0.780, t-test, 2 sided; Mean Difference (Final Values) = 3.21, 95% CI 2-sided [-20.3 to 26.7], Standard Error of Mean 11.4
Statistical Analysis 11: Comparison: Standard Implementation vs Facilitated Implementation; t-test of group differences on Role Clarity at 1 year; Test type: Superiority; p = 0.474, t-test, 2 sided; Mean Difference (Final Values) = 11.46, 95% CI 2-sided [-23.19 to 46.11], Standard Error of Mean 12.54
Statistical Analysis 12: Comparison: Standard Implementation vs Facilitated Implementation; t-test of group differences on Goals at 1 year; Test type: Superiority; p = 0.267, t-test, 2 sided; Mean Difference (Final Values) = 10.0, 95% CI 2-sided [-8.21 to 28.21], Standard Error of Mean 8.78

3. Secondary Outcome: Peer Fidelity Measure
Description: The Peer Fidelity Measure assesses: a) peer specialist services and b) peer specialist implementation. The first part has 5 domains of peer services critical to the VA's peer support model (e.g., being a role model that recovery is possible; share personal recovery story). The second has 7 domains of implementation factors shown to either help or hinder PS deployment (e.g., role clarity, support for PS at higher organizational levels, regular supervision). Each domain has 1-2 questions (responses ranging from 1= not at all through 5=Very much with higher scores indicating higher fidelity. Min Value=1 and Max value =5. The Peer Fidelity Measure will be administered to both Peer Specialists and their supervisors. Analyses looked at discrepancies (difference in difference) between Peer Specialists and their Supervisors at each time point. Min discrepancy score is -4 and Max discrepancy score is 4. (calculated as Peer Specialist minus Peer Supervisor score)
Time Frame: 6 months, 1 year
Population: 6 months and 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Implementation | Facilitated Implementation
Number analyzed (Participants) | 8 | 19
units on a scale
  Core Peer Specialist 6-moFunctions | 0.3 (0.3) | 0.7 (1.1)
  Collaborate-Promoting Health 6-mo | 0.2 (0.7) | 0.7 (1.2)
  Peer Specialist as Liaison 6-mo | -0.1 (1.2) | 1.1 (1.4)
  Provides Info on Services 6 mo | -0.1 (1.1) | 0.7 (0.8)
  Symptoms and Medications 6-mo | 0.2 (2.2) | 1.0 (2.0)
  Training and Preparation 6-mo | 0.1 (1.1) | 0.4 (1.6)
  Teams Integration and Relationships 6-mo | -0.4 (1.3) | 0.5 (1.5)
  Leadership Support 6-mo | 0.01 (1.2) | -0.2 (0.8)
  Fits to Experience and Needs 6-mo | -0.4 (1.6) | -0.4 (2.1)
  Role Clarity 6-mo | -0.3 (1.2) | 0.2 (1.3)
  Resources 6-mo | -0.1 (1.2) | 0.7 (1.6)
  Performance Reviews 6-mo | -0.1 (1.2) | -0.1 (2.3)
  Core PS functions 1-yr: number analyzed (Participants) | 2 | 10
  Core PS functions 1-yr | 0.7 (0.5) | -0.1 (0.41)
  Collaborate on Promoting Health 1 year: number analyzed (Participants) | 2 | 10
  Collaborate on Promoting Health 1 year | 0.7 (0.1) | -0.01 (0.6)
  Peer Specialist as Liaison 1 year: number analyzed (Participants) | 2 | 10
  Peer Specialist as Liaison 1 year | 0.8 (1.1) | -0.2 (0.6)
  provides info on services 1 year: number analyzed (Participants) | 2 | 10
  provides info on services 1 year | 0.0 (0.0) | -0.2 (0.5)
  Symptoms and Medication 1 year: number analyzed (Participants) | 2 | 10
  Symptoms and Medication 1 year | 0.8 (2.5) | -0.1 (2.1)
  Training and Preparation 1 year: number analyzed (Participants) | 2 | 10
  Training and Preparation 1 year | 0.5 (1.2) | -0.4 (1.1)
  Team Integration and relationships 1 year: number analyzed (Participants) | 2 | 10
  Team Integration and relationships 1 year | 1.1 (0.4) | -0.2 (0.5)
  Leadership Support 1 year: number analyzed (Participants) | 2 | 10
  Leadership Support 1 year | 2.5 (0.7) | 0.1 (1.1)
  Fit to experience and need 1 year: number analyzed (Participants) | 2 | 10
  Fit to experience and need 1 year | 0.0 (2.8) | -0.3 (0.8)
  Role Clarity 1 year: number analyzed (Participants) | 2 | 10
  Role Clarity 1 year | 1.3 (1.1) | -0.2 (0.9)
  Resources: number analyzed (Participants) | 2 | 10
  Resources | -0.5 (1.4) | -0.3 (0.5)
  Performance Review 1 year: number analyzed (Participants) | 2 | 10
  Performance Review 1 year | 0.8 (0.4) | -0.7 (2.2)
Statistical Analysis 1: Comparison: Standard Implementation vs Facilitated Implementation; t test comparison across groups on CORE PEER at 6 months; Test type: Superiority; p = 0.098, t-test, 2 sided; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [-0.09 to 1.00], Standard Error of Mean 0.38
Statistical Analysis 2: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on COLLABORATION at 6 months; Test type: Superiority; p = 0.282, t-test, 2 sided; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.43 to 1.43], Standard Error of Mean 1.1
Statistical Analysis 3: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on PEER SPECIALIST AS LIAISON at 6 months; Test type: Superiority; p = 0.06, t-test, 2 sided; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-0.05 to 2.29], Standard Error of Mean 0.56
Statistical Analysis 4: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on PROVIDES INFO ON SERVICES at 6 months; Test type: Superiority; p = 0.34, t-test, 2 sided; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [0.07 to 1.59], Standard Error of Mean 0.86
Statistical Analysis 5: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on Symptoms and Medication at 6-months; Test type: Superiority; p = 0.34, t-test, 2 sided; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [-0.94 to 2.62]
Statistical Analysis 6: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on Training and Preparation at 6-months; Test type: Superiority; p = 0.66, t-test, 2 sided; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-1.03 to 1.50], Standard Error of Mean 0.64
Statistical Analysis 7: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on Team Integration and Relationships at 6 Months; Test type: Superiority; p = 0.15, t-test, 2 sided; Mean Difference (Final Values) = 0.90, 95% CI 2-sided [-0.36 to 2.16], Standard Error of Mean 0.61
Statistical Analysis 8: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on Leadership at 6-months; Test type: Superiority; p = 0.59, t-test, 2 sided; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-1.01 to 0.59], Standard Error of Mean 0.39
Statistical Analysis 9: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on Fits to Experience at 6 months; Test type: Superiority; p = 0.95, t-test, 2 sided; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-1.77 to 1.68], Standard Error of Mean 0.84
Statistical Analysis 10: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on Role Clarity at 6 months; Test type: Superiority; p = 0.32, t-test, 2 sided; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [-0.58 to 1.68], Standard Error of Mean 0.55
Statistical Analysis 11: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across both groups on Resources at 6 months; Test type: Superiority; p = 0.27, t-test, 2 sided; Mean Difference (Final Values) = 0.72, 95% CI 2-sided [-0.60 to 2.04], Standard Error of Mean 0.64
Statistical Analysis 12: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on Performance Reviews at 6 months; Test type: Superiority; p = 0.93, t-test, 2 sided; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-1.71 to 1.85], Standard Error of Mean 0.86
Statistical Analysis 13: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on CORE PEER at 1 year; Test type: Superiority; p = 0.15, t-test, 2 sided; Mean Difference (Final Values) = -0.73, 95% CI 2-sided [-1.45 to -0.005], Standard Error of Mean 0.32
Statistical Analysis 14: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on Collaboration at 1 year; Test type: Superiority; p = 0.04, t-test, 2 sided; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.7 to 0.32], Standard Error of Mean 0.45
Statistical Analysis 15: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on Peer Specialists as Liaison at 1 year; Test type: Superiority; p = 0.08, t-test, 2 sided; Hazard Ratio, log = -0.95, 95% CI 2-sided [-2.07 to 0.17], Standard Error of Mean 0.50
Statistical Analysis 16: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on Provides Info on Services at 1 year; Test type: Superiority; p = 0.26, t-test, 2 sided; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.58 to 0.18], Standard Error of Mean 0.39
Statistical Analysis 17: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison between groups on Symptoms and Medication at 1 year; Test type: Superiority; p = 0.61, t-test, 2 sided; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-4.53 to 2.83], Standard Error of Mean 1.65
Statistical Analysis 18: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on Training and Preparation at 1 year; Test type: Superiority; p = 0.30, t-test, 2 sided; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-2.87 to 1.01], Standard Error of Mean 0.87
Statistical Analysis 19: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on Team Integration and Relationships at 1 year; Test type: Superiority; p = 0.004, t-test, 2 sided; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-2.08 to -0.52], Standard Error of Mean 0.35
Statistical Analysis 20: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on Leadership at 1 year; Test type: Superiority; p = 0.01, t-test, 2 sided; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-4.20 to -0.60], Standard Error of Mean 0.81
Statistical Analysis 21: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on Fits to Experience at 1 year; Test type: Superiority; p = 0.90, t-test, 2 sided; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-24.1 to 23.5], Standard Error of Mean 0.90
Statistical Analysis 22: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on Role Clarity at 1 year; Test type: Superiority; p = 0.06, t-test, 2 sided; Mean Difference (Final Values) = -1.45, 95% CI 2-sided [-3.02 to 0.12], Standard Error of Mean 0.70
Statistical Analysis 23: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison across groups on Resources at 1 year; Test type: Superiority; p = 0.71, t-test, 2 sided; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.97 to 1.37], Standard Error of Mean 0.53
Statistical Analysis 24: Comparison: Standard Implementation vs Facilitated Implementation; t-test comparison on Performance Reviews at 1 year; Test type: Superiority; p = 0.41, t-test, 2 sided; Mean Difference (Final Values) = -1.40, 95% CI 2-sided [-5.03 to 2.23], Standard Error of Mean 1.63

4. Secondary Outcome: The Satisfaction Index-Mental Health
Description: The Satisfaction Index-Mental Health is a 12-item, unidimensional measure of patient satisfaction with care. It has been used with Veteran populations and has been shown to be valid, reliable, and sensitive to change in a sample of Veterans with mental illnesses being treated in primary care settings. It will be administered to Veterans who receive care from the Peer Specialists involved in the project. Minimum score is 12 and the maximum score is 72; higher scores mean more satisfaction.
Time Frame: Baseline, 6 months, 1 year
Population: Veterans responding to survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Implementation | Facilitated Implementation
Number analyzed (Participants) | 194 | 221
units on a scale
  Baseline | 47.7 (12.1) | 51.3 (11.5)
  6-months: number analyzed (Participants) | 121 | 129
  6-months | 49.7 (12.7) | 52.3 (12.6)
  1-year: number analyzed (Participants) | 100 | 113
  1-year | 50.6 (13.0) | 51.2 (13.6)
Statistical Analysis 1: Comparison: Standard Implementation vs Facilitated Implementation; Group Comparison at Baseline; Test type: Superiority; p = 0.002, t-test, 2 sided — not adjusted for multiple comparisons; Mean Difference (Final Values) = 3.59, 95% CI 2-sided [1.29 to 5.88], Standard Error of Mean 1.17
Statistical Analysis 2: Comparison: Standard Implementation vs Facilitated Implementation; Group Comparison at 6 Months; Test type: Superiority; p = 0.10, t-test, 2 sided; Mean Difference (Final Values) = 2.62, 95% CI 2-sided [-0.54 to 5.78], Standard Error of Mean 1.60
Statistical Analysis 3: Comparison: Standard Implementation vs Facilitated Implementation; Group Comparison at 1 year; Test type: Superiority; p = 0.77, t-test, 2 sided; Mean Difference (Final Values) = 0.54, 95% CI 2-sided [-3.06 to 4.14], Standard Error of Mean 1.83

5. Secondary Outcome: Number of Unique Veterans Seen (Adjusted for Employment Period and Hours Worked Per Week)
Description: This adjusted workload variables took into consideration both the employment period (many PSs did not start immediately or may have left prior to the end of the 2 years) and weekly hours worked (varying from one hour to 40 hours per week). Visits during each PS's employment period were divided by the total number of hours worked, then multiplied by 40 to calculate adjusted values for operationalization above. Because this variable was significantly skewed, we used a log transformation to improve their distributional properties. Differences between intervention conditions were then compared with a series of Analyses of Covariance models with age, gender and race as covariates. Since these variables are measured at the PS level, the covariates were the average across the Veterans sesn by each PS (mean age, percent White and percent male). N's are number of Veterans
Time Frame: one year, across two years
Population: Unique Veteran encounters
Measure: Mean (Standard Deviation); unit: count of Veterans
Arm/Group | Standard Implementation | Facilitated Implementation
Number analyzed (Participants) | 899 | 1,484
count of Veterans
  1st year | 1.3 (1.3) | 4.8 (6.1)
  across both years | 5.8 (8.5) | 6.0 (5.8)
Statistical Analysis 1: Comparison: Standard Implementation vs Facilitated Implementation; Test type: Superiority; p = 0.02, t-test, 2 sided — p value for 1st year only; Mean Difference (Final Values) = 3.47, 95% CI 2-sided [0.56 to 6.38], Standard Error of Mean 1.56
Statistical Analysis 2: Comparison: Standard Implementation vs Facilitated Implementation; Test type: Superiority; p = 0.93, t-test, 2 sided; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-4.67 to 5.04], Standard Error of Mean 2.39

6. Secondary Outcome: Average Number of Visits Per Veteran Per Peer Specialist-Adjusted (Across Both Years)
Description: See Variable 5 above for details about adjustment. Since this variable this is a Veteran level variable, a General Linear Mixed Model (GSLMM) was used with PS specified as a random effect and Veteran age, race and gender.
  N's are number of Veterans
Time Frame: across both years
Population: Number of Visits per Veteran
Measure: Mean (Standard Deviation); unit: Count of Visits
Arm/Group | Standard Implementation | Facilitated Implementation
Number analyzed (Participants) | 899 | 1,484
Count of Visits | 2.2 (3.0) | 3.2 (5.6)
Statistical Analysis 1: Comparison: Standard Implementation vs Facilitated Implementation; Test type: Superiority; p = 0.0001, t-test, 2 sided; p value for 1st year; Mean Difference (Final Values) = 1.02, 95% CI 2-sided [0.68 to 1.37], Standard Error of Mean 0.20

7. Secondary Outcome: Average Total Number of Services Provided-Adjusted (First Year Only and Across Both Years)
Description: as for outcome 5
Time Frame: one year and across both years
Population: Services Provided by each Peer Specialist
Measure: Mean (Standard Deviation); unit: Count of services
Groups:
- Standard Implementation: Standard Implementation sites will receive written guidance and limited consultation by the in vestigators' team.
Arm/Group | Standard Implementation | Facilitated Implementation
Number analyzed (Participants) | 899 | 1,484
Count of services
  1st Year Only | 2.7 (2.7) | 8.4 (8.7)
  Across Both Years | 9.8 (8.7) | 12.4 (8.7)
Statistical Analysis 1: Comparison: Standard Implementation vs Facilitated Implementation; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Final Values) = 5.7, 95% CI 2-sided [1.46 to 9.96], Standard Error of Mean 2.26
Statistical Analysis 2: Comparison: Standard Implementation vs Facilitated Implementation; Test type: Superiority; p = 0.38, t-test, 2 sided; Mean Difference (Final Values) = 2.60, 95% CI 2-sided [-3.14 to 8.54], Standard Error of Mean 2.92

8. Secondary Outcome: Time to First Service
Description: This variable represents count of days from time study at each site started (baseline) until first service was delivered.
Time Frame: variable from baseline to time of first service delivered by Peer Specialists
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Standard Implementation | Facilitated Implementation
Number analyzed (Participants) | 16 | 21
Number of Days | 188.2 (123.4) | 88.7 (65.0)
Statistical Analysis 1: Comparison: Standard Implementation vs Facilitated Implementation; Test type: Superiority; p = 0.027, t-test, 2 sided; Mean Difference (Final Values) = -99.4, 95% CI 2-sided [-186.2 to -12.66], Standard Error of Mean 41.73

9. Secondary Outcome: Average Number of Visits Per Veteran Per Peer Specialist-Adjusted (First Year Only)
Description: as for outcome 6
Time Frame: 1st year only
Population: number of visits per Veteran
Measure: Mean (Standard Deviation); unit: Count of Visits
Arm/Group | Standard Implementation | Facilitated Implementation
Number analyzed (Participants) | 459 | 767
Count of Visits | 2.0 (2.1) | 2.6 (3.6)
Statistical Analysis 1: Comparison: Standard Implementation vs Facilitated Implementation; Test type: Superiority; p = 0.001, t-test, 2 sided; Mean Difference (Final Values) = 0.60, 95% CI 2-sided [0.28 to 0.92], Standard Error of Mean 0.18

ADVERSE EVENTS:
Time Frame: adverse events were not monitored or collected
Description: adverse events were not monitored or collected
Arm/Group | Standard Implementation | Facilitated Implementation
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
While the uploaded Study Protocol is in publication form, this represents the only written study protocol. Because the study was classified as non-research, there is no IRB protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT02732600/Prot_SAP_000.pdf